CLINICAL TRIAL: NCT05134883
Title: Effects of Hamstrings Flexibility After Proprioceptive Neuromuscular Facilitation Stretching Compared to Self-myofascial Release: a Randomized Controlled Trial
Brief Title: PNF Stretching Compared to SMR on Hamstrings
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Albert Pérez Bellmunt, Principal Investigator, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PNF_01
Record Dates: First submitted 2021-10-12; First posted 2021-11-26 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Sports Physical Therapy
Keywords: Stretching; Propioceptive neuromuscular facilitation; Hamstrings

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propioceptive neuromuscular facilitation (PNF) (Experimental): This group will undergo a PNF stretching on the hamstring muscles.
  Interventions: Other: PNF
- self myo-fascial release (SMR) (Active Comparator): This group will undergo a SMR stretching on the hamstring muscles.
  Interventions: Other: SMR

INTERVENTIONS:
Other: PNF — A PNF stretching protocol will be performed with each participant assuming a long sitting position on a plinth with the knee maintained as extended as possible. At this moment, the participant will be asked to perform a maximum isometric hamstring muscle contraction for 5 seconds followed by 5 seconds of relaxation and 20 seconds of stretching. The therapist will show the participant how to maintain this isometric contraction with the flexion of the hip and ankle. Each participant will undergo 4 repetitions of PNF stretching (30 seconds/rep).
  Arms: Propioceptive neuromuscular facilitation (PNF)
Other: SMR — For the application of self-myofascial release, the subjects will assume a long sitting position on a firm and even surface by placing the arms backward and transferring their body weight to their palms. The roller foam, applied bilaterally, will be placed under the hamstrings and slowly moved back and forth from the ischial tuberosity to the popliteal fossa by applying pressure for 2 minutes.
  Arms: self myo-fascial release (SMR)

SUMMARY:
The use of stretching techniques in the sports world is frequent and widely used for its many effects. One of the main benefits is the gain in flexibility, range of motion and facilitation of the sporting performance. Recently the use of self-myofascial release (SMR) has spread in sports practice both at elite and recreational level for its benefits being similar to those observed in stretching. The objective of the following study is to compare the results of the proprioceptive neuromuscular facilitation stretching with SMR on the hamstring muscle flexibility.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* hypermobility
* hamstring injury in the previous 6 months
* diagnosed orthopedic problems
* surgery in the lower limbs
* back pain
* spine surgery
* systemic or neurological disorders.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-10-05 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2022-01-30 (Estimated)

PRIMARY OUTCOMES:
Hamstring muscle flexibility (mm) | Change between baseline(immediately before intervention), mid-intervention (30 seconds after the start of the intervention) and post intervention (2 minutes after the start of the intervention)
  Evaluated with a modified sit-and-reach test (MSR). The participants sit on the floor with their lower limbs stretched out and together, their backs and hips are supported against the wall (90° hip flexion), and the soles of their feet are placed against the edge of a box. Participants then extended their arms forward, placing the same hand on top of the other with both hands facing down. During this, they keep their backs against the wall. They then reach forward, sliding their hands along the measuring scale as far as possible without bending their knees

SECONDARY OUTCOMES:
Discomfort sensation | Change between baseline(immediately before intervention), mid-intervention (30 seconds after start of intervention) and post intervention (2 minutes after the start of the intervention)
  Measured using the Borg rating of perceived exertion scale (RPE). The participants will be asked at the end of the intervention to give a number from 1 to 10, where 1 is the easiest and 10 the hardest.

CONTACTS AND LOCATIONS:
Overall Officials: Albert Pérez-Bellmunt, PhD, Principal Investigator — Universitat International Catalunya
Locations (1):
- Universitat Internacional Catalunya, Barcelona, Sant Cugat, Spain

REFERENCES:
- [Derived] Perez-Bellmunt A, Casasayas-Cos O, Ragazzi P, Rodriguez-Sanz J, Hidalgo-Garcia C, Canet-Vintro M, Caballero-Martinez I, Pacheco L, Lopez-de-Celis C. Foam Rolling vs. Proprioceptive Neuromuscular Facilitation Stretching in the Hamstring Flexibility of Amateur Athletes: Control Trials. Int J Environ Res Public Health. 2023 Jan 12;20(2):1439. doi: 10.3390/ijerph20021439. PMID 36674197